CLINICAL TRIAL: NCT04377815
Title: FORECAST Study: Finding Out if COVID-19 Infection Can be pREdicted by ChAnges in Smell and/or Taste
Brief Title: Finding Out if COVID-19 Infection Can be pREdicted by ChAnges in Smell and/or Taste
Acronym: FORECAST
Status: Completed | Type: Observational
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: 132311; 20/HRA/1879 (Other: Queen Square REC)
Record Dates: First submitted 2020-04-24; First posted 2020-05-06 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: COVID-19; Anosmia
Keywords: COVID-19; anosmia; taste
MeSH Terms: conditions — COVID-19; Anosmia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- General Public cohort: General Public
  Interventions: Other: General Public cohort
- Hospital cohort: Medical records of patients hospitalised due to COVID-19

INTERVENTIONS:
Other: General Public cohort — No intervention is being tested
  Other Names: Hospital cohort
  Groups: General Public cohort

SUMMARY:
The FORECAST Study is an observational cohort study looking at two cohorts of patients presenting with COVID-19: a general public cohort, aiming to investigate if new loss or reduced sense of smell and/or taste are early signs of COVID-19 and a hospital cohort, which will investigate if taste/smell changes can predict the clinical course of a COVID-19 infection.

DETAILED DESCRIPTION:
The FORECAST Study is an observational cohort study looking at two cohorts of patients presenting with COVID-19: a general public cohort, aiming to investigate if new loss or reduced sense of smell and/or taste are early signs of COVID-19 and a hospital cohort, which will investigate if taste/smell changes can predict the clinical course of a COVID-19 infection.

The main of objective of this study is to investigate whether loss/or reduced sense of smell and/or taste in the absence of fever and/or persistent cough are indicative of Coronavirus Infectious disease 2019 (COVID-19) infection. In addition, the study aims to investigate whether loss/or reduced sense of smell and/or taste precede the development of fever and persistent cough in people with COVID-19 infection and also whether loss of/reduced sense of smell and/or taste changes can be used to predict the clinical course of the disease.

General public FORECAST: Participants over the age of 18 will be sent a text message invite through participating GP practices' patient messaging systems. This will direct participants to a website (hosted by Dendrite Clinical Systems) where study subjects will find the participant information sheet, screening checks and consent form. Enrolled participants will complete an online questionnaire containing questions about smell and taste changes, as well as other symptoms of COVID-19. Participants will then be sent a near-patient rapid antibody test kit for COVID-19 to be undertaken only under medical supervision. Participants will be booked for a video conference appointment with either a doctor or nurse and the screening test will be performed under medical supervision. The outcome of the test will be documented, discussed with the patient and appropriate advice given. Four weeks after completing the first questionnaire participant will be sent an email and / or text message asking them to complete a second questionnaire.

This second questionnaire will contain questions about resolution of smell/taste symptoms and other symptoms of COVID-19. In case COVID-19 positive patients are subsequently admitted to hospital as a result of COVID-19, consent will be obtained to collect information on the outcome of the admission from discharge letter via GP. The data obtained will be analysed to determine if smell/taste symptoms alone are indicative of COVID-19 infection, whether smell/taste symptoms are early symptoms fo COVID-19 infection and whether smell/taste changes can be used to predict the clinical course of COVID-19 disease.

Hospital FORECAST: clinical records of patients admitted to University College London Hospital (UCLH) and the Whittington Hospital as a result of COVID-19 will be reviewed. The clinical notes of COVID-19 positive patients where absence or presence of smell/taste changes have been documented will be selected for review. Anonymised clinical data will be collected about symptoms on admission, the course of illness and outcomes. The study primary outcome will be to compare case fatility rate in COVID-19 postivite with documented history of loss/reduced sense of smell and/or taste compared to COVID-19 postive with documented history of no loss/reduced sense of smell and/or taste. The study will investigate whether loss/reduced sense of smell and/or taste can predict the course of illness and outcomes in COVID-19.

ELIGIBILITY:
General public FORECAST cohort: Participants will confirm their eligibility on the online form by confirming they meet the following inclusion and exclusion criteria:

Inclusion Criteria:

* Age over 18 years;
* Able to read and write English;
* Access to a computer or smartphone with internet access and ability to access video calling;
* Willingness to undertake a COVID-19 screening test;
* Willingness for their GP to be informed of their participation in the study.

Exclusion Criteria:

* Pre-existing smell or taste impairment of longer than 6 weeks duration;
* People lacking capacity.

Hospital FORECAST cohort: The patient records to be included in this part of the study will be selected by a healthcare professional based on the following inclusion and exclusion criteria

Inclusion Criteria:

* Admitted to hospital due to COVID-19 and documentation of either presense or absence of loss/reduced sense of smell and/or taste.

Exclusion Criteria:

* Changes in smell and/or taste either present or absent not documented.
* Admission due to other reason with later diagnosis of COVID-19 as an inpatient.
* Incomplete medical records.
* Patients with longstanding pre-existing smell and/or taste impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: General public FORECAST cohort
  Participating GP practices will send out text messages to potentially eligible patients registered with the practice inviting those who have noticed a recent (within the past 4 weeks) change (loss/decrease) in their sense of smell and/or taste to take part in a research study related to COVID-19 infection.
  Hospital FORECAST cohort
  For Hospital FORECAST, patients admitted with COVID-19 to UCLH and The Whittington Hospital will be identified through clinical coding. Their records will be reviewed by an appropriately qualified healthcare professional against the study's inclusion/exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 569 (Actual)
Dates: Start 2020-04-23 (Actual); Primary Completion 2020-05-14 (Actual); Study Completion 2020-06-24 (Actual)

PRIMARY OUTCOMES:
Percentage of people reporting changes in smell/taste | 4 weeks
  percentage of people who report loss/reduced sense of smell or taste
mortality rate | through study completion, an average of 1 year
  to compare the case mortality rate in COVID-19 patients who experienced smell/taste changes compared to mortality in those who did not experience smell/taste changes.

SECONDARY OUTCOMES:
Percentage of people with change in smell/taste before other symptoms | 4 weeks
  To identify the percentage of people who report changes in taste and/or smell before developing either fever or persistent cough who are positive for SARS-CoV-2 IgM and IgG
proportion of other COVID-19 linked symptoms in people with smell and/or taste change | 4 weeks
  To examine the proportion of other COVID-19 linked symptoms in people with smell and/or taste change who are positive positive for SARS-CoV-2 IgM and IgG who never develop fever and/or cough.
Percentage of people with persistent changes in smell and/or taste | 12 weeks
  To determine the percentage of people whose smell and/or taste symptoms persist for greater than 4 weeks in people who are positive for SARS-CoV-2 IgM and IgG
Percentage of hospitalisation | 12 weeks
  To determine the percentage of patients who report loss/decrease in sense of smell and/or taste changes before or in the absence of other symptoms of COVID-19, who are admitted to hospital with COVID-19
co-morbidities association | through study completion, an average of 1 year
  To investigate whether loss/reduced sense of smell and/or taste are associated with the course of illness and outcomes in COVID-19
prevalence of changes in smell/taste | through study completion, an average of 1 year
  Assessing the prevalence of previous loss/decrease in sense of smell and/or taste changes in patients admitted to secondary care with COVID-19 infection.
clinical outcomes | through study completion, an average of 1 year
  Correlating the presence of loss/decrease in sense of smell and/or taste changes to clinical outcomes including case fatality rate.

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - University College London Hospital, London
  - GP Practices, London

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Makaronidis J, Firman C, Magee CG, Mok J, Balogun N, Lechner M, Carnemolla A, Batterham RL. Distorted chemosensory perception and female sex associate with persistent smell and/or taste loss in people with SARS-CoV-2 antibodies: a community based cohort study investigating clinical course and resolution of acute smell and/or taste loss in people with and without SARS-CoV-2 antibodies in London, UK. BMC Infect Dis. 2021 Feb 25;21(1):221. doi: 10.1186/s12879-021-05927-w. PMID 33632171
- [Derived] Makaronidis J, Mok J, Balogun N, Magee CG, Omar RZ, Carnemolla A, Batterham RL. Seroprevalence of SARS-CoV-2 antibodies in people with an acute loss in their sense of smell and/or taste in a community-based population in London, UK: An observational cohort study. PLoS Med. 2020 Oct 1;17(10):e1003358. doi: 10.1371/journal.pmed.1003358. eCollection 2020 Oct. PMID 33001967